CLINICAL TRIAL: NCT03774147
Title: 24-hour Ambulatory Blood Pressure Monitoring in Patients With Blood Pressure Above Thresholds in General Practice
Acronym: MAPAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Burgundy (Other)
Collaborators: Association pour le Développement de la Recherche en Médecine Générale (ADRMG) (Unknown); Département de Médecine Générale de Dijon (DMG) (Unknown)
Responsible Party: Principal Investigator, Dr Claire ZABAWA, University senior registrar, University of Burgundy
Other Study IDs: 2014-A01536-41
Record Dates: First submitted 2018-12-04; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Hypertension; Blood Pressure Monitoring, Ambulatory; Primary Health Care
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 24-hour Ambulatory Blood Pressure Monitoring (ABPM)

SUMMARY:
High blood pressure (HBP) is a major modifiable cardiovascular risk factor which prevalence is gradually increasing. Reducing blood pressure (BP) significantly decreases cardiovascular morbi-mortality. Nevertheless, BP control remains insufficient: only 51% of French patients using antihypertensive drugs achieve the BP control targets.

HBP is mostly diagnosed and managed in primary care. Nevertheless, office BP measurements are unreliable for BP control and poorer predict target organ damage. Ambulatory BP measurements are recommended for HBP diagnosis and follow-up. 24-hour ambulatory blood pressure monitoring (ABPM) is the most cost-effective strategy. Its superiority has been demonstrated for HBP diagnosis and cardiovascular prognosis.

In France, ABPM is poorly available and little studied in primary care. Therefore, the investigators conducted a regional prospective study to analyze the feasibility and benefits of ABPM among primary care hypertensive patients in daily practice.

ELIGIBILITY:
Inclusion criteria:

* patients aged over 18 years
* with an office inclusion consultation systolic/diastolic BP≥ 140/90 mmHg
* able to understand French language and to consent to participate in the study

Exclusion criteria:

* patients aged < 18 years
* with conditions preventing technically adequate ABPM (chronic atrial fibrillation)
* with contraindications to ABPM (musculotendinous disease of the upper limb, past history of phlebitis of the upper limb or phlebitis in progress, past history of olecranon bursitis or bursitis in progress)
* with previous ABPM in the 12 months prior to the inclusion consultation
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-three general practitioners located in the four departments of the Burgundy region and practising in seven different health structures were recruited on a voluntary basis.
  Primary care patients with an office high blood pressure were included, whatever their reason for consultation, medical past history or ongoing treatment
Sampling Method: Probability Sample
Enrollment: 1067 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of white-coat hypertension | at the time of ABPM, up to 30 days after the inclusion consultation
  Proportion of patients with normotension in ABPM (daytime systolic/diastolic BP< 135/85 mmHg AND/OR nighttime BP< 120/70 mmHg AND/OR 24-hour BP< 130/80 mmHg) among the patients with primary care office measured BP≥ 140/90 mmHg
Prevalence of nocturnal hypertension | at the time of ABPM, up to 30 days after the inclusion consultation
  Proportion of patients with nocturnal high blood pressure in ABPM (nighttime systolic/diastolic BP> 120/70 mmHg) among the patients with primary care office measured BP≥ 140/90 mmHg
Prevalence of diurnal hypertension | at the time of ABPM, up to 30 days after the inclusion consultation
  Proportion of patients with diurnal high blood pressure in ABPM (daytime systolic/diastolic BP> 135/85 mmHg) among the patients with primary care office measured BP≥ 140/90 mmHg
Prevalence of 24-hour hypertension | at the time of ABPM, up to 30 days after the inclusion consultation
  Proportion of patients with 24-hour high blood pressure in ABPM (24-hour systolic/diastolic BP> 130/80 mmHg) among the patients with primary care office measured BP≥ 140/90 mmHg

SECONDARY OUTCOMES:
Dipping | at the time of ABPM, up to 30 days after the inclusion consultation
  Proportion of nighttime mean BP fall, compared to daytime mean BP
ABPM acceptability | at the time of ABPM, up to 30 days after the inclusion consultation
  Number of patients who have undergone/completed the ABPM
ABPM validity | at the time of ABPM, up to 30 days after the inclusion consultation
  Number of patients who have had an invalid ABPM according to the criteria of the European society of cardiology
ABPM side effects | at the time of ABPM, up to 30 days after the inclusion consultation
  Number of major side effects
Deprivation among hypertensive patients | at the time of ABPM, up to 30 days after the inclusion consultation
  Deprivation status of hypertensive primary care patients, according to the French Assessment of deprivation in Health Examination Centers' (EPICES) score (deprivation if EPICES score> 30)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Groupements des Professionnels de Santé du Pays Beaunois, Beaune
  - Maison Universitaire de Santé et de Soins Primaires, Chenôve
  - Cabinet de médecine générale, Garchizy
  - Maison de santé de Terre Pleine, Guillon
  - Maison de Santé Pluridisciplinaire, Montret
  - Groupement des Professionnels de Santé de l'Auxois Sud, Pouilly-en-Auxois
  - Maison de santé de l'Esplanade, Tournus

IPD SHARING:
Plan to Share IPD: No